CLINICAL TRIAL: NCT01588535
Title: Phase 2, Multicenter, Placebo-controlled, Double-masked, Randomized Study to Demonstrate Reliability and Validity of FAECC Scale (Modified FLACC) to Evaluate Relief of Pain in Subjects With Acute Otitis Media Aged >/=2 Months to <5 Years
Brief Title: Study of FAECC Scale (Modified FLACC) to Evaluate Ear Pain in Children With Acute Otitis Media
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AR01.004
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-03

CONDITIONS: Pain; Otitis Media
Keywords: pain; pain measurement; ear, middle; otitis media
MeSH Terms: conditions — Pain; Otitis Media | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- benzocaine solution (Active Comparator): ear drops
  Interventions: Drug: benzocaine
- Placebo (Placebo Comparator): ear drops
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: benzocaine — benzocaine 10 mg/mL, five drops in affected ear canal each hour as needed
  Other Names: Arbor otic; AR01
  Arms: benzocaine solution
Drug: placebo — placebo solution, five drops in affected ear canal each hour as needed
  Arms: Placebo

SUMMARY:
This study is to assess the reliability and validity of the FAECC scale to evaluate pain associated with acute otitis media in children aged 2 months to 5 years.

DETAILED DESCRIPTION:
to assess the reliability and validity of the FAECC pain scale tool in children aged 2 months to 5 years with acute otitis media given AR01 or placebo

ELIGIBILITY:
Inclusion Criteria:

* The patient has age in the interval 2 months ≤ age < 5.00 years, signs and symptoms of AOM, and moderate to severe pain (current episode ≤ 2 weeks duration). Moderate to severe pain is defined as a score of > or = 4 (on a scale of 0 - 10) for the FAECC scale as assessed by the primary assessor.
* The patient's parent/guardian must have read and signed the written informed consent prior to study participation.
* The patient is normally active and otherwise judged to be in good health on the basis of medical history and limited physical examination.

Exclusion Criteria:

* Patient has perforated tympanic membrane, history of a perforated tympanic membrane in the last 6 months, or if a perforated tympanic membrane could not be ruled out by speculum examination, impedance testing tympanometry, pneumatic otoscopy, or Valsalva maneuver. Patients who are subsequently diagnosed with a perforated membrane during treatment are to be discontinued immediately. Patients with tympanostomy tubes are not allowed.
* Patient has acute or chronic otitis externa.
* Patient has chronic otitis media (current episode ≥ 2 weeks).
* Patient has seborrheic dermatitis involving the affected external ear canal or pinna.
* Patient has received any otic topical or systemic antibiotic within 14 days prior to study entry (topical or systemic antibiotics for acne will be allowed on a chronic basis for subjects who have been on a stable dose for at least 14 days prior to entry).
* Patient has received any topical drying agent or over-the-counter therapy for otitis media within 36 hours prior to enrollment.
* Patient has fever ≤ 102.0 F (oral or equivalent).
* Patient has known hypersensitivity to the study drug or similar compounds including any of the inactive ingredients.
* Patient is receiving medication on a chronic basis for pain (including steroidal or non steroidal anti-inflammatory drugs) and has not been on a stable dose for at least 1 month prior to entry into the study.
* Patient has clinically significant mental illness (to be determined by the Investigator).
* Patient has been exposed to any investigational agent within 30 days prior to study entry.
* Patient has been previously enrolled in this study.
* Patient or caregiver (parent/guardian) has a condition the Investigator believes will interfere with the ability to provide consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk.
* Patient has a glucose 6-phosphate dehydrogenase deficiency or is taking concomitant medications associated with methemoglobinemia (such as nitrates or nitrites; aniline dyes; or medications, including lidocaine, prilocaine, phenazopyridine hydrochloride [Pyridium], and others).
* Patient demonstrates clinical signs of anemia. The absolute amount of deoxygenated or abnormal hemoglobin (rather than its percentage) is required for cyanosis to be clinically evident. Patients with moderate-to-severe anemia may not appear cyanotic, even with elevated percentages of deoxygenated or abnormal hemoglobin.
* Patient has congenital (i.e., hereditary) methemoglobinemia.
* Patient has a recent history of acute gastroenteritis within 14 days prior to study entry. An association between methemoglobinemia and acute gastroenteritis in infants has been noted in several studies and may be due to acidosis from stool bicarbonate loss impairing the already immature function of the methemoglobin reductase system in these young patients.

Ages: 2 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Consistency of primary assessor and caregiver FAECC scores using Pearson's correlation coefficient | up to 120 minutes after first dose and Day 4

SECONDARY OUTCOMES:
reduction in pain scores from predose to each post-dose time point | up to 120 minutes after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Downey, MD, Study Director — Arbor Pharmaceuticals, Inc.
Locations (15):
- United States (15):
  - Nda Baptist Clinic, Jonesboro, Arkansas
  - COMMUNITY Medical Research, Miami Beach, Florida
  - The Iowa Clinic, Pc, West Des Moines, Iowa
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Prairie Fields Family Medicine/Clinical Research Advantage, Fremont, Nebraska
  - Clinical Research Center, Las Vegas, Nevada
  - Odyssey Research, Fargo, North Dakota
  - ACCESS CLINICAL TRIALS, Inc. / Centennial Medical Center, Clarksville, Tennessee
  - DiscoveReseach, Inc., Bryan, Texas
  - Research Across America, Carrollton, Texas
  - Research Across America, Dallas, Texas
  - Dm Clinical Research, Tomball, Texas
  - Foothill Family Clinic, Salt Lake City, Utah
  - FIRSTMED, Salt Lake City, Utah
  - Jordon River Family Medicine, South Jordan, Utah